CLINICAL TRIAL: NCT06226376
Title: The Effects of EXOPULSE Mollii Suit on Fibromyalgia Syndrome in Patients With Fibromyalgia (EXOFIB 2): A Sham Controlled Randomized Double-Blind Trial
Brief Title: Mollii Suit and Fibromyalgia (EXOFIB 2)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheikh Shakhbout Medical City (Other)
Responsible Party: Principal Investigator, Naji Joseph Riachi, Principal Investigator, Sheikh Shakhbout Medical City
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: EXOFIB2
Record Dates: First submitted 2024-01-17; First posted 2024-01-26 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Fibromyalgia; Rheumatic Diseases; Muscular Diseases; Neuromuscular Diseases; Nervous System Diseases
MeSH Terms: conditions — Fibromyalgia; Rheumatic Diseases; Muscular Diseases; Neuromuscular Diseases; Nervous System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXOPULSE Mollii Suit Stimulation Active. (Active Comparator): This will be the EXOPULSE Mollii Suit Active Stimulation. Stimulation will go on for 60 minutes while control unit is on for 60 minutes.
  Interventions: Device: EXOPULSE Mollii Suit Stimulation
- EXOPULSE Mollii Suit Stimulation Sham. (Sham Comparator): This will be the EXOPULSE Mollii Suit Sham Stimulation. Stimulation will go on for 1 minute then it turns off while the control unit will remain on for total of 60 minutes
  Interventions: Device: EXOPULSE Mollii Suit Stimulation

INTERVENTIONS:
Device: EXOPULSE Mollii Suit Stimulation — We designed a randomized sham controlled double-blind trial to demonstrate the improvement of pain, quality of life, fatigue and mood in adult patients with fibromyalgia following a 2-week intervention of "active" versus "sham" Exopulse Mollii suit. A 2-week washout period should be enough to prevent a potential carry over effect. After this phase (phase 1), a second open label phase (phase 2) will be proposed for patients to understand the effects of Exopulse Mollii suit employed for 4 weeks (7 sessions per week) on the studied outcomes.

SUMMARY:
The goal of this clinical trial is to demonstrate the improvement of fibromyalgia syndrome obtained following active stimulation compared to sham, with diminished functional disability and improved health status using Exopulse Molli suit stimulation. The main questions it aims to answer are:

Evaluation of pain, fatigue, mood and quality of life changes observed after active stimulation in comparison to sham.

Improvement of fibromyalgia syndrome as per the Fibromyalgia Impact Questionnaire (FIQ)

Study subjects will participate in:

A randomized sham controlled double-blind trial to demonstrate the improvement of pain, quality of life, fatigue and mood in adult patients with fibromyalgia following a 2-week intervention of "active" versus "sham" Exopulse Mollii suit. A 2-week washout period should be enough to prevent a potential carry over effect. After this phase (phase 1), a second open label phase (phase 2) will be proposed for patients to understand the effects of Exopulse Mollii suit employed for 4 weeks (7 sessions per week) on the studied outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 75 years, with a definite diagnosis of fibromyalgia according to the American College of Rheumatology (ACR) 2010 criteria, set for at least one month.
* Patients should be able to understand verbal instructions.

Exclusion Criteria:

* Patient with VAS < 4
* Patient included in another research protocol during the study period
* Patient unable to undergo medical monitor for the study purposes due to geographical or social reasons
* Patient with contraindication to wearing Exopulse Mollii suit (e.g., cardiac stimulator, a ventriculoperitoneal shunt, intrathecal baclofen pump, pregnancy, and/or body mass index above 35 kg/m2)
* Patient with other somatic or psychiatric diagnoses other than anxiety and depression (e.g., arrhythmias, uncontrolled epilepsy, other diseases causing osteoarticular and muscular pain)
* Any change in the pharmacological therapy in the last three months
* Introduction of a medical device other than Exopulse Mollii suit during the study period
* Patient under juridical protection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2025-03-24 (Actual); Study Completion 2025-05-24 (Actual)

PRIMARY OUTCOMES:
Fibromyalgia Impact Questionnaire (FIQ) | This to be assessed at baseline, then at week 2, week 4, week 6, week 8 and week 12.
  It is an 11-item scale that assesses health status and functional disability by exploring the impact of fibromyalgia on work, wellbeing, fatigue, sleep, stiffness, anxiety, and depression. FIQ scores can range from 0 to 100, with higher scores reflecting worse health status. Scores could be used to classify fibromyalgia as mild (scores: 0-38), moderate (scores: 39-58), and severe (scores: 59-100)

SECONDARY OUTCOMES:
Brief Pain Inventory (BPI) | This to be assessed at baseline, then at week 2, week 4, week 6, week 8 and week 12.
  will be used to assess pain severity (4 items) and pain interference (7 items). BPI items are rated on a 10-point scale running from 0 (no pain/does not interfere) to 10 (pain as bad as the participant can imagine/interferes completely).
Pain Catastrophizing Scale (PCS) | This to be assessed at baseline, then at week 2, week 4, week 6, week 8 and week 12.
  Pain Catastrophizing Scale (PCS) will be employed, which is a valid and reliable scale that includes 13 items assessing the presence and severity of feelings or thoughts that emerge when experiencing pain. Each item is rated on a 5-point Likert scale ranging from 0 (not at all) to 4 (all the time). It is possible to calculate a total and three subscale scores (i.e., helplessness, magnification, and rumination)
Quality of life as per the Short Form 36 Health Survey (SF-36) | This to be assessed at baseline, then at week 2, week 4, week 6, week 8 and week 12.
  It is a generic survey that contains 36 items which assess the quality of life and yield eight dimensions: physical functioning, physical role, emotional role, bodily pain, general health, vitality, social functioning, and mental health. The score of each dimension ranges from 0 to 100, with higher scales implying better health status.
Visual Analogue Scale for Pain | This to be assessed at baseline, then at week 2, week 4, week 6, week 8 and week 12.
  Pain will be measured using a visual analog score from 0 to 10, 0 being no pain, to 10 being the worst possible pain.
Visual Analogue Scale for Fatigue | This to be assessed at baseline, then at week 2, week 4, week 6, week 8 and week 12.
  Fatigue will be measured using a visual analog score from 0 to 10, 0 being no fatigue, to 10 being the worst possible fatigue
Hospital Anxiety and Depression Scale (HADS) | This to be assessed at baseline, then at week 2, week 4, week 6, week 8 and week 12.
  It is a 14-item generic scale with good psychometric properties and consists of seven items assessing anxiety and seven others assessing depression. Scores can range from 0 to 21 on each subscale, with higher scores indicating worse symptomatology.
Clinical Global Impression (CGI) | This to be assessed at week 2, week 6 and week 12.
  Evaluation of overall Clinical improvement will be done using the 7-point Clinical Global Impression (CGI). Patient will fill a questionnaire that will address their clinical situation as follows:
  Very much improved. Much improved. Slightly improved. No change. Slightly worse Much worse. Very much worse The score will range from 1-7, 1 being the best clinical outcome and 7 the worst.

CONTACTS AND LOCATIONS:
Locations (1):
- SSMC, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Annemans L, Le Lay K, Taieb C. Societal and patient burden of fibromyalgia syndrome. Pharmacoeconomics. 2009;27(7):547-59. doi: 10.2165/11313650-000000000-00000. PMID 19663526
- [Background] Bengtsson A, Henriksson KG. The muscle in fibromyalgia--a review of Swedish studies. J Rheumatol Suppl. 1989 Nov;19:144-9. PMID 2691674
- [Background] Bocerean C, Dupret E. A validation study of the Hospital Anxiety and Depression Scale (HADS) in a large sample of French employees. BMC Psychiatry. 2014 Dec 16;14:354. doi: 10.1186/s12888-014-0354-0. PMID 25511175
- [Background] Burckhardt CS, Clark SR, Bennett RM. The fibromyalgia impact questionnaire: development and validation. J Rheumatol. 1991 May;18(5):728-33. PMID 1865419
- [Background] Burwinkle T, Robinson JP, Turk DC. Fear of movement: factor structure of the tampa scale of kinesiophobia in patients with fibromyalgia syndrome. J Pain. 2005 Jun;6(6):384-91. doi: 10.1016/j.jpain.2005.01.355. PMID 15943960
- [Background] Busner J, Targum SD. The clinical global impressions scale: applying a research tool in clinical practice. Psychiatry (Edgmont). 2007 Jul;4(7):28-37. PMID 20526405
- [Background] Campbell WI, Lewis S. Visual analogue measurement of pain. Ulster Med J. 1990 Oct;59(2):149-54. PMID 2278111
- [Background] Cleeland CS, Ryan KM. Pain assessment: global use of the Brief Pain Inventory. Ann Acad Med Singap. 1994 Mar;23(2):129-38. PMID 8080219
- [Background] Coskun Benlidayi I. The effectiveness and safety of electrotherapy in the management of fibromyalgia. Rheumatol Int. 2020 Oct;40(10):1571-1580. doi: 10.1007/s00296-020-04618-0. Epub 2020 Jun 10. PMID 32524302
- [Background] Da Silva TFG, Suda EY, Marçulo CA, Paes FHS, Pinheiro GT. Comparison of transcutaneous electrical nerve stimulation and hydrotherapy effects on pain, flexibility and quality of life in patients with fibromyalgia [Comparação dos efeitos da estimulação elétrica nervosa transcutânea e da hidroterapia na dor, flexibilidade e qualidade de vida de pacientes com fibromialgia]. Fisioterapia e Pesquisa 2008;15:118-24.
- [Background] Dailey DL, Rakel BA, Vance CGT, Liebano RE, Amrit AS, Bush HM, Lee KS, Lee JE, Sluka KA. Transcutaneous electrical nerve stimulation reduces pain, fatigue and hyperalgesia while restoring central inhibition in primary fibromyalgia. Pain. 2013 Nov;154(11):2554-2562. doi: 10.1016/j.pain.2013.07.043. Epub 2013 Jul 27. PMID 23900134
- [Background] Dailey DL, Vance CGT, Rakel BA, Zimmerman MB, Embree J, Merriwether EN, Geasland KM, Chimenti R, Williams JM, Golchha M, Crofford LJ, Sluka KA. Transcutaneous Electrical Nerve Stimulation Reduces Movement-Evoked Pain and Fatigue: A Randomized, Controlled Trial. Arthritis Rheumatol. 2020 May;72(5):824-836. doi: 10.1002/art.41170. Epub 2020 Mar 18. PMID 31738014
- [Background] Drewes AM, Andreasen A, Schroder HD, Hogsaa B, Jennum P. Pathology of skeletal muscle in fibromyalgia: a histo-immuno-chemical and ultrastructural study. Br J Rheumatol. 1993 Jun;32(6):479-83. doi: 10.1093/rheumatology/32.6.479. PMID 8508284
- [Background] Elvin A, Siosteen AK, Nilsson A, Kosek E. Decreased muscle blood flow in fibromyalgia patients during standardised muscle exercise: a contrast media enhanced colour Doppler study. Eur J Pain. 2006 Feb;10(2):137-44. doi: 10.1016/j.ejpain.2005.02.001. PMID 16310717
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] French DJ, Noël M, Vigneau F, French JA, Cyr CP, Evans RT. [PCS-CF: A French-language, French-Canadian adaptation of the Pain Catastrophizing Scale]. Canadian Journal of Behavioural Science. 2005;37:181-192.
- [Background] Ghavidel-Parsa B, Bidari A, Amir Maafi A, Ghalebaghi B. The Iceberg Nature of Fibromyalgia Burden: The Clinical and Economic Aspects. Korean J Pain. 2015 Jul;28(3):169-76. doi: 10.3344/kjp.2015.28.3.169. Epub 2015 Jul 1. PMID 26175876
- [Background] Johnson MI, Claydon LS, Herbison GP, Jones G, Paley CA. Transcutaneous electrical nerve stimulation (TENS) for fibromyalgia in adults. Cochrane Database Syst Rev. 2017 Oct 9;10(10):CD012172. doi: 10.1002/14651858.CD012172.pub2. PMID 28990665
- [Background] Kahl C, Cleland J. Visual Analogue Scale, Numeric Rating Scale and the McGill Pain Quesitonniare: An Overview of Psychometric Properties. Phys Ther. 2005;10:123.
- [Background] Kim SK, Kim SH, Lee CK, Lee HS, Lee SH, Park YB, Park HJ, Son MJ, Lee SS. Effect of fibromyalgia syndrome on the health-related quality of life and economic burden in Korea. Rheumatology (Oxford). 2013 Feb;52(2):311-20. doi: 10.1093/rheumatology/kes255. Epub 2012 Sep 28. PMID 23024016
- [Background] Macfarlane GJ, Kronisch C, Dean LE, Atzeni F, Hauser W, Fluss E, Choy E, Kosek E, Amris K, Branco J, Dincer F, Leino-Arjas P, Longley K, McCarthy GM, Makri S, Perrot S, Sarzi-Puttini P, Taylor A, Jones GT. EULAR revised recommendations for the management of fibromyalgia. Ann Rheum Dis. 2017 Feb;76(2):318-328. doi: 10.1136/annrheumdis-2016-209724. Epub 2016 Jul 4. PMID 27377815
- [Background] Marques AP, Assumpcao A, Matsutani LA, Pereira CA, Lage L. Pain in fibromyalgia and discrimination power of the instruments: Visual Analog Scale, Dolorimetry and the McGill Pain Questionnaire. Acta Reumatol Port. 2008 Jul-Sep;33(3):345-51. PMID 18846013
- [Background] Okifuji A, Hare BD. Management of fibromyalgia syndrome: review of evidence. Pain Ther. 2013 Dec;2(2):87-104. doi: 10.1007/s40122-013-0016-9. Epub 2013 Sep 21. PMID 25135147
- [Background] Park JH, Phothimat P, Oates CT, Hernanz-Schulman M, Olsen NJ. Use of P-31 magnetic resonance spectroscopy to detect metabolic abnormalities in muscles of patients with fibromyalgia. Arthritis Rheum. 1998 Mar;41(3):406-13. doi: 10.1002/1529-0131(199803)41:33.0.CO;2-L. PMID 9506567
- [Background] Perneger TV, Leplege A, Etter JF, Rougemont A. Validation of a French-language version of the MOS 36-Item Short Form Health Survey (SF-36) in young healthy adults. J Clin Epidemiol. 1995 Aug;48(8):1051-60. doi: 10.1016/0895-4356(94)00227-h. PMID 7775992
- [Background] Perrot S, Dumont D, Guillemin F, Pouchot J, Coste J; French Group for Quality of Life Research. Quality of life in women with fibromyalgia syndrome: validation of the QIF, the French version of the fibromyalgia impact questionnaire. J Rheumatol. 2003 May;30(5):1054-9. PMID 12734906
- [Background] Queiroz LP. Worldwide epidemiology of fibromyalgia. Curr Pain Headache Rep. 2013 Aug;17(8):356. doi: 10.1007/s11916-013-0356-5. PMID 23801009
- [Background] Riachi N, Khazen G, Ahdab R, Jörgen S. Pain reducing properties of the Mollii suit on adults with chronic pain syndromes. J. Neurol. Sci. 2019;405:138-139
- [Background] Schaefer C, Chandran A, Hufstader M, Baik R, McNett M, Goldenberg D, Gerwin R, Zlateva G. The comparative burden of mild, moderate and severe fibromyalgia: results from a cross-sectional survey in the United States. Health Qual Life Outcomes. 2011 Aug 22;9:71. doi: 10.1186/1477-7525-9-71. PMID 21859448
- [Background] Schmidt-Wilcke T, Clauw DJ. Fibromyalgia: from pathophysiology to therapy. Nat Rev Rheumatol. 2011 Jul 19;7(9):518-27. doi: 10.1038/nrrheum.2011.98. PMID 21769128
- [Background] Schmidt-Wilcke T, Diers M. New Insights into the Pathophysiology and Treatment of Fibromyalgia. Biomedicines. 2017 May 13;5(2):22. doi: 10.3390/biomedicines5020022. PMID 28536365
- [Background] Sprott H, Rzanny R, Reichenbach JR, Kaiser WA, Hein G, Stein G. 31P magnetic resonance spectroscopy in fibromyalgic muscle. Rheumatology (Oxford). 2000 Oct;39(10):1121-5. doi: 10.1093/rheumatology/39.10.1121. PMID 11035133
- [Background] Steffen TM, Hacker TA, Mollinger L. Age- and gender-related test performance in community-dwelling elderly people: Six-Minute Walk Test, Berg Balance Scale, Timed Up & Go Test, and gait speeds. Phys Ther. 2002 Feb;82(2):128-37. doi: 10.1093/ptj/82.2.128. PMID 11856064
- [Background] Sullivan MJ, Bishop SR, Pivik J. The Pain Catastrophizing Scale: Development and validation. Psychol Assess. 1995;7:524-532.
- [Background] Taylor SJ, Steer M, Ashe SC, Furness PJ, Haywood-Small S, Lawson K. Patients' perspective of the effectiveness and acceptability of pharmacological and non-pharmacological treatments of fibromyalgia. Scand J Pain. 2019 Jan 28;19(1):167-181. doi: 10.1515/sjpain-2018-0116. PMID 30315738
- [Background] Ware JE Jr, Snow KK, Kosinski M, Gandek B. SF-36 health survey: manual and interpretation guide. Boston: The Health Institute, New England Medical Center; 1993.
- [Background] Winkelmann A, Perrot S, Schaefer C, Ryan K, Chandran A, Sadosky A, Zlateva G. Impact of fibromyalgia severity on health economic costs: results from a European cross-sectional study. Appl Health Econ Health Policy. 2011 Mar 1;9(2):125-36. doi: 10.2165/11535250-000000000-00000. PMID 21332254
- [Background] Wolfe F, Brahler E, Hinz A, Hauser W. Fibromyalgia prevalence, somatic symptom reporting, and the dimensionality of polysymptomatic distress: results from a survey of the general population. Arthritis Care Res (Hoboken). 2013 May;65(5):777-85. doi: 10.1002/acr.21931. PMID 23424058
- [Background] Wolfe F, Walitt BT, Hauser W. What is fibromyalgia, how is it diagnosed, and what does it really mean? Arthritis Care Res (Hoboken). 2014 Jul;66(7):969-71. doi: 10.1002/acr.22207. No abstract available. PMID 24127234
- [Background] Wolfe F, Clauw DJ, Fitzcharles MA, Goldenberg DL, Katz RS, Mease P, Russell AS, Russell IJ, Winfield JB, Yunus MB. The American College of Rheumatology preliminary diagnostic criteria for fibromyalgia and measurement of symptom severity. Arthritis Care Res (Hoboken). 2010 May;62(5):600-10. doi: 10.1002/acr.20140. PMID 20461783